CLINICAL TRIAL: NCT00096343
Title: A Phase II Trial of Pre-Operative Taxol and Carboplatin in Women With Newly Diagnosed Locally Advanced Operable Breast Cancer
Brief Title: Paclitaxel and Carboplatin in Treating Women Who Are Undergoing Surgery for Newly Diagnosed, Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisle Nabell, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000377728; UAB-0137
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; invasive lobular breast carcinoma; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Inflammatory Breast Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel IV followed by Carboplatin IV (Experimental): paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before surgery may shrink the tumor so that it can be removed. Combining paclitaxel with carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with carboplatin works in treating women who are undergoing surgery for newly diagnosed, locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical and pathological response in women with newly diagnosed, locally advanced operable breast cancer treated with neoadjuvant chemotherapy comprising paclitaxel and carboplatin.
* Evaluate specific biomarkers for prognostic value and as markers for response/resistance in patients treated with this regimen.
* Determine the tolerability and toxicity of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients with non-palpable lymph nodes undergo sentinel lymph node biopsy within 4 weeks before beginning neoadjuvant chemotherapy.

All patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo lumpectomy or modified radical mastectomy. Patients with a positive sentinel lymph node biopsy or palpable axillary adenopathy undergo axillary lymph node dissection. All patients undergoing lumpectomy or mastectomy with high-risk disease also undergo radiotherapy.

Patients refusing lumpectomy or mastectomy due to persistence of disease may undergo core needle biopsy.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive ductal carcinoma or invasive lobular carcinoma of the breast meeting the following stage criteria:

  * T2, T3, or T4a-c
  * N0-2
  * M0
* Inflammatory breast cancer (stage IIIB) allowed
* Measurable disease by mammogram or ultrasound
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.2 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No comorbid medical condition that would preclude study participation
* No comorbid infection that would preclude study participation
* No clinically significant peripheral neuropathy (> grade 1)
* No prior significant allergic reaction to drugs containing Cremophor, such as teniposide, cyclosporine, or vitamin K
* No dementia or altered mental status that would prohibit understanding of informed consent
* No other primary malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic growth factors

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* At least 3 weeks since prior surgery

Other

* No other concurrent anticancer drugs

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-10; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Determine the clinical and pathological response in women with newly diagnosed, locally advanced operable breast cancer treated with neoadjuvant chemotherapy comprising paclitaxel and carboplatin | baseline to 18 months

SECONDARY OUTCOMES:
Evaluate specific biomarkers for prognostic value and as markers for response/resistance in patients treated with this regimen | baseline through 18 months
Determine the tolerability and toxicity of this regimen in these patients. | baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisle M. Nabell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States